CLINICAL TRIAL: NCT01884532
Title: Cross-Sectional, Multi-Center Evaluation of 6 Year Metal Ion Trends for ASR-XL Total Hip Replacement System
Brief Title: ASR-XL Metal-on-Metal 522 Post-Market Surveillance Study
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 11012
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-05

CONDITIONS: Adverse Local Tissue Reaction; Total Hip Arthroplasty
Keywords: Adverse Local Tissue Reaction; Metal Ions; Serum; Whole Blood; Metal-on-Metal; Total Hip Arthroplasty; ASR-XL Metal-on-Metal; Revised ASR-XL Metal-on-Metal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and serum samples are retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 2 year post-op: Patients that underwent an ASR-XL Metal-on-Metal (MoM) total hip replacement (THR)and at the time of enrollment, based on their date of surgery, were 2 years post-operative. Alternatively, these are patients who have had their ASR-XL Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: ASR-XL Metal-on-Metal
- 3 year post-op: Patients that underwent an ASR-XL Metal-on-Metal (MoM) total hip replacement (THR)and at the time of enrollment, based on their date of surgery, were 3 years post-operative. Alternatively, these are patients who have had their ASR-XL Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: ASR-XL Metal-on-Metal
- 4 year post-op: Patients that underwent an ASR-XL Metal-on-Metal (MoM) total hip replacement (THR)and at the time of enrollment, based on their date of surgery, were 4 years post-operative. Alternatively, these are patients who have had their ASR-XL Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: ASR-XL Metal-on-Metal
- 5 year post-op: Patients that underwent an ASR-XL Metal-on-Metal (MoM) total hip replacement (THR)and at the time of enrollment, based on their date of surgery, were 5 years post-operative. Alternatively, these are patients who have had their ASR-XL Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: ASR-XL Metal-on-Metal
- 6 year post-op: Patients that underwent an ASR-XL Metal-on-Metal (MoM) total hip replacement (THR)and at the time of enrollment, based on their date of surgery, were 6 years post-operative. Alternatively, these are patients who have had their ASR-XL Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: ASR-XL Metal-on-Metal

INTERVENTIONS:
Device: ASR-XL Metal-on-Metal — All patients that are post-operative will have undergone total hip arthroplasty with the ASR-XL Metal-on-Metal device.
  Other Names: ASR-XL; ASR-XL MoM

SUMMARY:
The purpose of this clinical study is to evaluate blood metal ion levels as a function of time of implantation for the ASR-XL MoM system.

ELIGIBILITY:
Inclusion Criteria:

1. Able to (or capable of) provide written, voluntary consent to participate in the clinical investigation,
2. Is willing and able to return for all protocol defined clinic visits,
3. Subject has (or had, if previously revised) a combination of the following implants in the study hip:

   1. ASR-XL cup or ASR 300 cup
   2. XL femoral head
   3. ASR-XL tapered sleeve adapter
   4. One of the following stems

   i. S-ROM ii. Corail iii. Tri-Lock iv. AML v. Summit vi. Prodigy vii. C-Stem AMT
4. Subject has high quality films available for review that were taken within 12 months of primary surgery of the following views:

   1. Standing AP-Pelvis
   2. Standing AP-Proximal Femur (if this view is not available but the AP-Pelvis shows the entire implant and greater trochanter, that is also acceptable)
   3. Lauenstien Lateral Proximal Femur (Lateral-femur).

Exclusion Criteria:

1. The subject refuses to allow their medical records to be inspected by the Sponsor, representatives of the Sponsor, the medical office staff and/or representatives from the FDA
2. The implanted hip components in the study hip (exclusive of cement), are not all DePuy components
3. The femoral component is the ASR hemi or some other hemi device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have undergone a total hip arthroplasty with the ASR-XL Metal-on-Metal device that are currently 2 to 6 years post-operative.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Chromium serum ion level across time intervals | Pre-operatively through 6 years
  To compare the chromium serum ion levels in the patient population from pre-operatively through 6 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (2 through 6 years) will be a different cohort of patients. Notes: Pre-operative values are being collected via a separate protocol. There is no 1 year data available for this product due its withdrawal from the market.
Change in Chromium whole blood ion level across time intervals | Pre-operatively through 6 years
  To compare the chromium whole blood ion levels in the patient population from pre-operatively through 6 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (2 through 6 years) will be a different cohort of patients. Notes: Pre-operative values are being collected via a separate protocol. There is no 1 year data available for this product due its withdrawal from the market.
Change in Cobalt serum ion level across time intervals | Pre-operatively through 6 years
  To compare the cobalt serum ion levels in the patient population from pre-operatively through 6 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (2 through 6 years) will be a different cohort of patients. Notes: Pre-operative values are being collected via a separate protocol. There is no 1 year data available for this product due its withdrawal from the market.
Change in Cobalt whole blood ion level across time intervals | Pre-operatively through 6 years
  To compare the cobalt whole blood ion levels in the patient population from pre-operatively through 6 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (2 through 6 years) will be a different cohort of patients. Notes: Pre-operative values are being collected via a separate protocol. There is no 1 year data available for this product due its withdrawal from the market.

SECONDARY OUTCOMES:
Poolability of data across stem types | Pre-operatively through 6 years post-operatively
  Within each of the primary analyses, the poolability of the data across stem types will be confirmed with a 2-way ANOVA model in which both time interval and stem type are independent variables. Note: Pre-operative data is being collected via a separate protocol.
Incidence of adverse local tissue reaction (ALTR) | Pre-operatively through 6 years post-operatively
  To determine trends in the incidence of ALTR over time.
Implant survivorship | Through 6 years post-operatively
  To determine implant survivorship, where an implant is considered to be surviving when none of the total hip replacement (THR)system components have been removed or replaced, so that the original system with metal-on-metal (MoM) articulating surfaces remains intact. Implant survivorship will be analyzed in two ways: 1) for all revisions (for any reason)and 2) for revisions due to ALTR.
To identify the incidence of ALTR among unrevised subjects | Through 6 years post-operatively
  To identify the incidence of ALTR among unrevised subjects through physical examination and imaging.
Ion levels among revised subjects | Pre-operatively through 6 years post-operatively
  To compare cobalt and chromium ion level (prior to revision) vs. baseline for subjects who are revised. Note: Pre-operative levels are being obtained via a separate protocol.
Harris Hip and HOOS analysis for pain, function and total score | Through 6 years post-operatively
  To identify the incidence of pain or functional symptoms among unrevised subjects with a Harris Hip and HOOS evaluation. To compare cobalt and chromium ion levels for unrevised subject who are exhibiting pain or functional symptoms vs. unrevised subject who are not exhibiting pain or functional symptoms.
To determine the association of adverse events with elevated ion levels | Through 6 years post-operatively
  To investigate the association of adverse events with elevated cobalt and chromium ion levels. For each respective adverse event, to compare cobalt and chromium ion levels for subjects who have vs. subjects who have not exhibited the adverse event. For each respective adverse event category, to present summary statistics of cobalt and chromium ion levels for subjects who have vs. subjects who have not exhibited the adverse event, stratified by post-op time cohort.
Trending | Through 6 years post-operatively
  Trends (over time since initial implant) will be evaluated for : 1) revisions (survivorship), 2) adverse events, 3) pain or functional symptoms (via Harris Hip and HOOS evaluations), 4) incidence of ALTR in unrevised subjects
Patient history and demographics and association with outcomes | Throughout 6 years post-operatively
  Patient demographic and subject history will be evaluated for association with: 1) higher metal ion levels and 2) risk of revision
Modes and causes of implant failure | Through 6 years post-operatively
  To evaluate modes and causes of implant failure based on an analysis of reasonably available explanted retrieved devices.
Metal ion levels and association with reason for revision | Through 6 years post-operatively
  To compare cobalt and chromium levels across the different reasons for revision.
Comparison of metal ion levels across subjects with vs. without ALTR | Through 6 years post-operatively
  Cobalt and chromium ion levels will be compared for unrevised subjects who were not diagnosed with an ALTR vs. unrevised subjects who were diagnosed with an ALTR.
Ion level vs. baseline for ALTR subjects | Through 6 years post-operatively
  To compare cobalt and chromium ion level vs. baseline for subjects who are diagnosed with ALTR. Note: Baseline measurements are being captured via a separate protocol.
Ion level change from first measurement for ALTR subjects | Through 6 years post-operatively
  Cobalt and chromium ion levels will be compared from first measurement to the time of revision (prior to revision) or the time of last follow-up visit in the study, whichever comes first, for subjects who are diagnosed with an ALTR.

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Panozzo, BS, Study Director — DePuy Synthes Joint Reconstruction
Locations (7):
- United States (7):
  - Fort Collins, Colorado
  - Glenview, Illinois
  - Rockford, Illinois
  - Las Vegas, Nevada
  - Durham, North Carolina
  - Cincinnatti, Ohio
  - Austin, Texas